CLINICAL TRIAL: NCT04910828
Title: Effect of High and Low Glycemic Index Foods on Post Meal Pulse and Blood Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, David Jenkins, Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REB 20-114
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Heart Rate; Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Common foods of varying glycemic indices (Experimental): Common foods of varying glycemic indices
  Interventions: Other: Common foods of varying glycemic indices

INTERVENTIONS:
Other: Common foods of varying glycemic indices — Examples of foods of varying glycemic index to be tested include bread, rice, breakfast cereals, starchy vegetables, legumes, fruit and dairy products.

SUMMARY:
The aim of this study is to test high and low glycemic index foods in healthy adult volunteers and determine the effects on post meal pulse and blood pressure. Foods will be consumed before 8am after an overnight fast (10-12 hours) over a 10-15 minute period. Pulse and BP (where equipment is available) measurements will be taken 6 times at 5 min intervals before eating, and twice every 15 min thereafter for the following 2h. We will recruit between 30 to 40 students and 10 to 20 older adults to assess the effect of age, in cohorts of 10.

DETAILED DESCRIPTION:
STUDY OBJECTIVE

The aim of this study is to test high and low glycemic index foods in healthy volunteers and determine the effects on post meal pulse and blood pressure.

METHODS

Participants: 30 to 40 students and 10 to 20 older adults (>60 years) will be recruited.

Inclusion:

-Healthy adult volunteers

Exclusion:

-Serious health condition preventing participants from eating 50g of "available" carbohydrates as a test breakfast. For example: 1) food intolerances or allergies to common foods; 2) gastrointestinal conditions requiring medical treatment (Crohn's, ulcerative colitis) and a special diet; 3) bariatric surgery.

Recruitment Study participants will be recruited from those who have contacted us and showed interest in working with our group as well as colleagues who show interest in this project. The study coordinator will obtain consent by telephone and confirm by email.

Study Design Fifty of the original 65 carbohydrate foods, as used in the 1981 AJCN (American Journal Of Clinical Nutrition) glycemic index paper, that established the first comprehensive values for the glycemic index of foods, will be fed to healthy volunteers as 50g carbohydrate portions as was done for the original GI testing. Foods will be consumed before 8am after an overnight fast (10-12 hours) over a 10-15 minute period. Pulse and BP (where equipment is available) measurements will be taken 6 times at 5 min intervals before eating, and twice every 15 min thereafter for the following 2h. Participants will be asked to test at least 10 (or more as they wish) foods on separate days. The minimum duration for their participation will therefore be 10 days but not necessarily consecutively.

Sample Size We will recruit between 30 to 40 students and 10 to 20 older adults to assess the effect of age, in cohorts of 10, and to have the flexibility for volunteers to do less foods but still have a wide range of foods on which to obtain a tachycardia or hypotension index.

Procedures Prior to starting the study, they will be asked to complete a medical questionnaire sent to them by email and return it to the study coordinator for review. Participants will either come to the Risk Factor Modification Centre at St. Michael's Hospital if pandemic restrictions allow, or will carry out the testing by themselves at home. Tests will be carried out after an overnight fast. Participants will sit quietly for 15 minutes and then repeat pulse (and BP with the Omron or other monitor if available) measurements 6 x at 5 min intervals or until measurements are consistent for 3 consecutive readings.

The test meal breakfast will then be eaten over 10-15 minutes, with 2 further pulse measurements taken at 15 minute intervals for the following 2h after the start of breakfast.

Throughout, participants will be asked to remain seated and emotionally uninvolved with their environment. Pulse can be counted for 30 seconds to ensure concentration (and x by 2 for the minute value). Written work, answering emails etc. can be undertaken providing the timing of pulse measurements does not induce stress. The first 2h are crucial in this respect.

Study Intervention/Breakfasts Participants will be given a list of 10 foods (including white bread to be used as the standard), and their weights and method of preparation. They will acquire these common foods themselves. If they have no scales available, they will portion the foods using common measures and the values with which they will be provided. Cooking instructions will also be provided where necessary. Food portions should be measured out the night before and left in the refrigerator overnight.

Foods will be consumed plain or with a set weight of fat (e.g. butter or margarine) or protein (cottage cheese or tofu). A beverage of their choice (tea or coffee) will also be taken with either cow or soy milk or water. The quantities should be constant across all test breakfasts and the total volume of the beverage should be 300 ml.

Foods A list of foods, portion sizes, preparation instructions and order in which to eat them will be provided prior to the start of the study.

Study test diary form Forms on which to record timing and study details (cooking instructions for lentils, pasta etc.) will be provided for each test.

Scales and measuring jugs Where possible participants should ensure that they have electronic scales with wall plugs that are in gram weights and also jugs with ml volume calibrations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers

Exclusion Criteria:

* Serious health condition preventing participants from eating 50g of "available" carbohydrates as a test breakfast. For example: 1) food intolerances or allergies to common foods; 2) gastrointestinal conditions requiring medical treatment (Crohn's, ulcerative colitis) and a special diet; 3) bariatric surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Heart Rate (pulse) | 2 hours following consumption of food
  Heart Rate (pulse)
Blood pressure | 2 hours following consumption of food
  Blood pressure